CLINICAL TRIAL: NCT03494868
Title: Preoperative Oral Carbohydrate Drink for Elective Cesarean Delivery and the Effect on Insulin Sensitivity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: need additional funding
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Emily E. Sharpe, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-009567
Record Dates: First submitted 2018-04-04; First posted 2018-04-11 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Insulin Sensitivity
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fasting (No Intervention): Fasting prior to elective cesarean section delivery (standard of care)
- Carbohydrate Drink (Experimental): Subjects will drink 2 carbohydrate drinks prior to elective cesarean section delivery
  Interventions: Dietary Supplement: Carbohydrate Drink

INTERVENTIONS:
Dietary Supplement: Carbohydrate Drink — 2 - 12 oz drinks
  Other Names: Clearfast Preop Drink
  Arms: Carbohydrate Drink

SUMMARY:
Preoperative fasting and surgery can cause metabolic stress and insulin resistance. Oral carbohydrate loading has been shown to attenuate the development of insulin resistance in the non-pregnant population undergoing many different types of surgery. Pregnant women have an increase in insulin resistance and therefore may further benefit from a preoperative carbohydrate load prior to cesarean delivery. Although woman in the UK receive a carbohydrate drink prior to elective cesarean delivery, the metabolic effects of these drinks on the mother and neonate have not been evaluated.

DETAILED DESCRIPTION:
Preoperative fasting and surgery can cause metabolic stress and insulin resistance. Perioperative insulin resistance results in hyperglycemia which can lead to increased infectious complications, morbidity, and mortality.2,3 Significant research has occurred in the non-pregnant population utilizing preoperative oral carbohydrate loading to attenuate the development of insulin resistance. In a recent meta-analysis, Awad and colleagues 2 found that a preoperative carbohydrate drink may be associated with reduced length of stay and a reduction in postoperative insulin resistance in patients undergoing major abdominal surgery.

Approximately 1.3 million women undergo cesarean delivery (CD) annually in the United States. 4 CD is the most common inpatient surgery in the United States. In the UK, there are recommendations to implement enhanced recovery after obstetric surgery. Implementation of enhanced recovery supports the National Health Service Quality, Innovation, Productivity, and Prevention programme with the aim of improving quality of care while reducing costs. As part of the enhanced recovery pathway, pregnant women are receiving a preoperative carbohydrate drink. There is a paucity of research looking at the metabolic effects of this carbohydrate load in the pregnant woman and her neonate.

ELIGIBILITY:
Inclusion:

* ASA physical status II-III women presenting for scheduled, elective cesarean delivery under neuraxial anesthesia
* Singleton gestation at term (37-42 weeks)
* Ages 18-50

Exclusion:

* Preexisting diabetes (Gestational diabetes, Type I DM, Type II DM)
* Taking insulin-sensitizing or other medications known to influence glucose or fatty acid metabolism.
* Kidney, heart, or liver disease. Severe lipid disorders.
* History of bariatric surgery
* Pre-pregnancy BMI >40
* Prolonged period of time (>4 hours) between ingestion of carbohydrate drink and surgery
* Four or more repeat cesarean sections

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2025-04-29 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
Oral glucose tolerance test | 24 hours postoperatively
  glucose, insulin

CONTACTS AND LOCATIONS:
Overall Officials: Emily E Sharpe, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials